CLINICAL TRIAL: NCT00013507
Title: Effects of Functional Incidental Training in VA NHCU Residents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: E2226R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Aging
Keywords: Frail; FIT; transfer; continence; ambulation; balance; fall risk; strength,endurance
MeSH Terms: interventions — Accidental Falls

INTERVENTIONS:
Procedure: Falls

SUMMARY:
This research on Functional Incidental Training ( FIT) primarily involves women residing in community nursing homes. It is an individualized rehabilitative protocol intended to improve mobility, endurance, strength and continence in frail, older, functionally impaired and disabled veterans.

Objectives of the project are as follows:

1) Test the effects of FIT on transfer ability, continence, ambulation/mobility, balance and fall risk, strength, and endurance; 2) Determine the characteristics of NHCU residents who respond to FIT; 3)Identify the most sensitive outcome measures related to FIT; and 4) Determine the labor costs of FIT relative to usual care.

DETAILED DESCRIPTION:
This research on Functional Incidental Training ( FIT) primarily involves women in community nursing homes.

Objectives:

1. test the effects of FIT on functions such as transfer ability, continence, ambulation/mobility,balance and fall risk, strength, and endurance; 2. determine the characteristics of NHCU residents who respond to FIT; 3. identify the most sensitive outcome measures related to FIT; and 4. determine the labor costs of FIT relative to usual care.

. The intervention is an individualized rehabilitative protocol intended to improve mobility, endurance, strength and continence in frail, older, functionally impaired and disabled veterans in VA nursing home care units(NHCUs).The design is a multi-site cross-over design, to be carried out in five NHCUs (Atlanta, Durham, Salisbury, Augusta, Tuscaloosa) over about eight months in each site. About 24 residents will be recruited in each NHCU: 12 each will be randomized to initial intervention and control for 8 wks and evaluated; the controls will then receive the intervention and vice versa for another 8 wks with another evaluation. Patients are seen 4x a day for FIT activities, including walking/using wheel chair, prompted toileting, strengthening exercises. Outcome measures will be made in a blinded manner by Project Manager.

ELIGIBILITY:
Functionally impaired elderly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1999-01; Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D., Asst. Director — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Victoria Mongiardo, Program Analyst — Department of Veterans Affairs, Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Decatur, Decatur, Georgia, United States